CLINICAL TRIAL: NCT07138716
Title: Application Study of 68Ga-DOTA-CCK-FS PET/CT in Medullary Thyroid Carcinoma (MTC) and Various Other Tumors With Positive Expression of Cholecystokinin-2 Receptor (CCK-2R)
Brief Title: Research on the Application of 68Ga-DOTA-CCK-FS PET/CT in MTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luo Yaping (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor-Investigator, Luo Yaping, Medical Doctor (M.D.), Chief Physician, Professor, Assistant Director, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CCK-2R
Record Dates: First submitted 2025-05-07; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Medullary Thyroid Carcinoma
Keywords: MTC; CCK-2R; PET/CT
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 68Ga-DOTA-CCK-FS and 68Ga-DOTA-TATE PET/CT imaging (Other): For the patients with neuroendocrine neoplasm. Intravenous administration of 1.8-2.2 MBq/kg (0.05-0.06 mCi/kg) of each radiotracer within one week. For 68Ga-DOTA-CCK-FS, imaging begins 60±5 minutes post-injection to evaluate cholecystokinin receptor (CCK-R) expression, while 68Ga-DOTA-TATE scanning starts at 45-60 minutes post-injection for somatostatin receptor (SSTR) assessment, both using a time-of-flight PET/CT system with low-dose CT (120 kVp, 30-50 mAs) for attenuation correction followed by whole-body PET acquisition (2-3 min/bed position). Images are reconstructed using OSEM algorithms
  Interventions: Diagnostic Test: 68Ga-DOTA-CCK-FS PET/CT
- 68Ga-DOTA-CCK-FS and 18F-FDG PET/CT imaging (Other): For the patients with non-neuroendocrine neoplasm. 68Ga-DOTA-CCK-FS PET/CT was perfomed 60±5 minutes post-injection of 1.8-2.2 MBq/kg (0.05-0.06 mCi/kg) tracer. The 18F-FDG PET/CT imaging protocol requires patients to fast for at least 6 hours and maintain blood glucose levels <150-200 mg/dL prior to intravenous administration of 3.7-5.2 MBq/kg (0.1-0.14 mCi/kg) of 18F-FDG. After a 60±5 minute uptake period , imaging is performed on a time-of-flight PET/CT system (2-3 minutes per bed position, covering skull base to mid-thigh).
  Interventions: Diagnostic Test: 68Ga-DOTA-CCK-FS PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-DOTA-CCK-FS PET/CT — For 68Ga-DOTA-CCK-FS, imaging begins 60±5 minutes post-injection to evaluate cholecystokinin receptor (CCK-R) expression, using a time-of-flight PET/CT system with low-dose CT (120 kVp, 30-50 mAs) for attenuation correction followed by whole-body PET acquisition (2-3 min/bed position). Images are reconstructed using OSEM algorithms.

SUMMARY:
This study explores the clinical application of 68Ga-DOTA-CCK-FS PET/CT in detecting cholecystokinin-2 receptor (CCK-2R)-positive tumors, particularly medullary thyroid cancer (MTC) and other malignancies. Led by Prof. Luo Yaping (PUMCH Nuclear Medicine) and Prof. Liu Zhibo (Peking University, radiochemistry expert), the trial will enroll 30-40 patients to compare 68Ga-DOTA-CCK-FS imaging with standard PET/CT (e.g., 18F-FDG or 68Ga-DOTATATE). The novel tracer shows higher tumor uptake and retention in preclinical studies, potentially improving diagnosis and treatment guidance for aggressive, CCK-2R-expressing cancers. The study leverages PUMCH's Class IV Radioactive Drug License for advanced radiopharmaceutical development. Risks are minimal (diagnostic radiation dose only), and participants receive free imaging assessments. Results aim to refine precision diagnostics for MTC and related tumors.

DETAILED DESCRIPTION:
This clinical study investigates the diagnostic potential of 68Ga-DOTA-CCK-FS PET/CT, a novel radiopharmaceutical targeting the cholecystokinin-2 receptor (CCK-2R), in patients with medullary thyroid carcinoma (MTC) and other CCK-2R-expressing tumors. The research is led by Prof. Luo Yaping, Chief Physician at Peking Union Medical College Hospital (PUMCH), in collaboration with Prof. Liu Zhibo, a radiochemistry expert from Peking University. The trial will enroll 30-40 eligible patients with confirmed or suspected MTC (based on histopathology, elevated calcitonin/CEA levels, or MEN2 family history) or other CCK-2R-positive malignancies. Each participant will undergo 68Ga-DOTA-CCK-FS PET/CT, with comparative imaging (either 18F-FDG PET/CT for non-neuroendocrine tumors or 68Ga-DOTATATE PET/CT for neuroendocrine tumors) performed within 2 weeks. The study focuses on evaluating the tracer's sensitivity, specificity, and tumor-targeting efficiency through both visual and quantitative analyses (e.g., SUV measurements). Preclinical data suggest 68Ga-DOTA-CCK-FS offers superior tumor uptake and retention compared to existing probes, potentially enabling earlier detection and better therapeutic stratification for MTC, which often presents with aggressive metastasis and limited treatment options. PUMCH's Class IV Radioactive Drug License allows in-house production of this investigational tracer, addressing unmet clinical needs. Safety monitoring includes tracking minor injection-site reactions or radiation exposure (equivalent to a standard abdominal CT). Participants benefit from free advanced imaging and contribute to refining precision diagnostics for CCK-2R-driven cancers. Results may pave the way for future theranostic applications (e.g., 177Lu-labeled CCK-2R therapy).

ELIGIBILITY:
Inclusion Criteria:

1. Age not limited (male or female).
2. Diagnosis:Confirmed or suspected medullary thyroid carcinoma (MTC) based on:

   Fine-needle aspiration (FNA) cytology/histopathology, or Elevated serum calcitonin/CEA with thyroid nodule(s), or Clinical/hereditary suspicion (e.g., MEN2 syndrome), or Other histologically confirmed CCK-2R-positive tumors (e.g., neuroendocrine tumors, gastric/ovarian cancers).
3. Performance Status: Life expectancy ≥12 weeks.
4. Contraception: Willingness to use effective birth control (if applicable).
5. Consent: Signed informed consent and compliance with follow-up.

Exclusion Criteria:

1. Severe hepatic/renal dysfunction (e.g., ALT/AST >3×ULN, Cr >2.0 mg/dL).
2. Pregnancy/lactation or planned pregnancy during the study.
3. Inability to lie still for PET/CT (e.g., severe claustrophobia).
4. Concurrent conditions compromising study safety (investigator's judgment).

*Note: CCK-2R positivity may be confirmed via prior immunohistochemistry (if available) or inferred from tumor type (e.g., MTC).*

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance | through study completion, an average of 1 year
  Diagnostic performance of 68Ga-DOTA-CCK-FS PET/CT in detecting CCK-2R-positive tumors, as measured by sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy using histopathology or clinical follow-up as the reference standard.

SECONDARY OUTCOMES:
Comparative efficacy | through study completion, an average of 1 year
  Comparative efficacy of 68Ga-DOTA-CCK-FS PET/CT versus standard imaging (18F-FDG PET/CT for non-neuroendocrine tumors or 68Ga-DOTATATE PET/CT for neuroendocrine tumors) in:
  Tumor detection rate (number and location of lesions)
  Target-to-background ratio (TBR) based on SUVmax (tumor vs. liver/blood pool/muscle)
Correlation | through study completion, an average of 1 year
  Correlation between 68Ga-DOTA-CCK-FS uptake (SUVmax/SUVpeak) and Serum tumor markers (e.g., calcitonin, CEA for MTC); Tumor differentiation status (if histopathology is available)
Safety profile | through study completion, an average of 1 year
  Safety profile of 68Ga-DOTA-CCK-FS, assessed by Incidence of adverse events (AEs) related to tracer administration and Radiation dosimetry estimates

OTHER OUTCOMES:
Exploratory Outcomes | through study completion, an average of 1 year
  Potential utility of 68Ga-DOTA-CCK-FS PET/CT for:
  Staging/restaging of MTC and other CCK-2R-positive tumors Predicting eligibility for future peptide receptor radionuclide therapy (PRRT) Inter-reader agreement in image interpretation (kappa statistics)

CONTACTS AND LOCATIONS:
Overall Officials: Yaping LUO, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Due to patient privacy regulations and institutional policies, individual participant data (IPD) from this study will not be publicly available. The data contain sensitive clinical and genetic information that could compromise participant confidentiality. Additionally, Chinese data protection laws and hospital ethical guidelines restrict the open sharing of identifiable medical data.
  However, aggregated results (e.g., group-level imaging findings, statistical analyses) will be published in peer-reviewed journals. Researchers may request limited, anonymized datasets for collaborative purposes, subject to approval by the Peking Union Medical College Hospital (PUMCH) Ethics Committee and compliance with data transfer agreements.